CLINICAL TRIAL: NCT03685643
Title: Study Protocol for a Peer-led Web-based Intervention to Promote Safe Usage of Dating Applications Amongst Young Adults: A Cluster Randomized Controlled Trial
Brief Title: Study Proposal for Web Based Intervention to Promote the Safe Usage of Dating Applications in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09160275; HKUCTR-2512 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Sex, Unsafe; Adolescent Behavior; Behavior, Sex
Keywords: Peer-led, dating applications, young adults, sexual behavior
MeSH Terms: conditions — Unsafe Sex; Adolescent Behavior; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Dating application topic (Experimental): The intervention will consist of four short videos with points of discussion, a scenario game, and a risk assessment tool regarding dating application usage.
  Interventions: Behavioral: Intervention - Dating application topic
- Control - Health and exercise topic (Placebo Comparator): The control will consist of four short videos with discussion points and an interaction game regarding exercise and healthy living tips.
  Interventions: Behavioral: Control - Health and exercise topic

INTERVENTIONS:
Behavioral: Intervention - Dating application topic — The intervention will consist of multimedia content to promote the safe usage of dating applications and raise awareness of the risks associated with dating application usage. The intervention will be delivered one-time in a classroom setting.
  Arms: Intervention - Dating application topic
Behavioral: Control - Health and exercise topic — The placebo control will consist of multimedia content regarding exercise and healthy living. It will be delivered once-time in a classroom setting.
  Arms: Control - Health and exercise topic

SUMMARY:
This study will evaluate the effectiveness of a program in promoting the safe usage of dating applications amongst young adults in Hong Kong. One group will receive the program regarding dating applications and the other group will receive a placebo program regarding health and exercise.

DETAILED DESCRIPTION:
Dating applications are a popular platform to meet new people; however, they have been associated with risks such as unsafe sexual behavior and privacy concerns in young adults.

The study design is an open-labeled cluster randomized controlled trial with an intervention and a placebo control arm. The intervention group will receive a web-based intervention developed through focus group discussions, crowdsourcing contest, and a Peer-Vetted Creative Production (PVCP) workshop comprising of four short videos, a risk assessment tool, and a scenario game. The control group will receive a web-based resource with similar multimedia elements on health and exercise.

Based on the Information, Motivation, and Behavioral Skills (IMB) Model, the primary outcome of this study is self-efficacy in using dating applications measured by the General Self Efficacy Scale. Secondary outcomes include change in attitudes regarding risk perception measured by the Risk Propensity Scale and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 17-27 years old
* Able to read and understand Chinese

Exclusion Criteria:

* Have a physical impediment (e.g. blindness) to prevent them from accessing the content

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 578 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wong, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Caritas Institute of Community Education, Hong Kong
  - Vocational Training Council (VTC), Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data will include baseline demographics, dating application usage and behavior, and the primary and secondary outcomes.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 6 months after study completion.
Access Criteria: Data access requests will be reviewed by an external review panel.

REFERENCES:
- [Derived] Wong WC, Sun WH, Chia SMC, Tucker JD, Mak WP, Song L, Choi KWY, Lau STH, Wan EYF. Effectiveness of a Peer-Led Web-Based Intervention to Improve General Self-Efficacy in Using Dating Apps Among Young Adults: Randomized Clustered Trial. J Med Internet Res. 2020 Oct 30;22(10):e16378. doi: 10.2196/16378. PMID 33124987
- [Derived] Lau STH, Choi KWY, Chen J, Mak WP, Yeung HKCA, Tucker J, Wong WC. Study protocol for a peer-led web-based intervention to promote safe usage of dating applications among young adults: a cluster randomized controlled trial. Trials. 2019 Feb 6;20(1):102. doi: 10.1186/s13063-018-3167-5. PMID 30728064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 578 eligible participants (290 in the intervention and 288 in the control) participated in the study.
Groups:
- Intervention: The intervention materials were developed with high peer engagement and included four short videos, an interactive scenario game and a risk assessment tool.
- Control: An existing website promoting physical activities and healthy living was served as a control.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 290 | 288
Completed | 276 | 266
Not Completed | 14 | 22
Not completed — Lost to Follow-up | 14 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 276 | 266 | 542
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 19.83 (1.9) | 19.88 (1.8) | 19.86 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 179 | 318
  Male | 137 | 87 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 276 | 266 | 542
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 276 | 266 | 542
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 276 | 266 | 542
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 250 | 240 | 490
  Others (gay, lesbian or bisexual) | 26 | 26 | 52
Relationship Status [Count of Participants; unit: Participants]
  Single | 183 | 170 | 353
  Others (Dating, marriage or cohabitating) | 93 | 96 | 189
Types of housing [Count of Participants; unit: Participants]
  Private Apartment | 107 | 101 | 208
  Public housing estates | 104 | 82 | 186
  Subsided housing | 34 | 39 | 73
  Student Hostel | 19 | 29 | 48
  Villiages | 7 | 15 | 22
  Short interim | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Self Efficacy: This Will be Measured by the General Self Efficacy Scale
Description: The primary outcome will be the self-efficacy on the safe usage of dating. applications among young adults in Hong Kong. This will be measured by the General Self Efficacy Scale. The General Self Efficacy Scale is a 10-item scale (with 4 level Likert scale ranging from "not true at all" to "exactly true") measuring one's self-belief in completing certain tasks or overcoming difficulties. The total score is calculated by finding the sum of all items with the total score ranging between 10 and 40, with a higher score indicating a higher level of self efficacy.
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention - Dating Application Topic | Control - Health and Exercise Topic
Number analyzed (Participants) | 290 | 288
Score on a scale | 24.26 (5.48) | 22.30 (4.69)
Statistical Analysis 1: Comparison: Intervention - Dating Application Topic vs Control - Health and Exercise Topic; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Risk Taking Tendencies Will be Measured by the The Risk Propensity Scale.
Description: Participants' risk taking tendencies will be measured by the The Risk Propensity Scale. It is a 9-item scale measuring general risk-taking tendencies. Each item is rated on a 9 level Likert scale (ranging from "totally disagree" to "totally agree") with the final score ranging from 1-9. A higher score indicates higher risk-taking tendencies.
Time Frame: 8 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention - Dating Application Topic | Control - Health and Exercise Topic
Number analyzed (Participants) | 290 | 288
Score on a scale | 5.42 (1.23) | 5.59 (1.15)
Statistical Analysis 1: Comparison: Intervention - Dating Application Topic vs Control - Health and Exercise Topic; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Depression Symptoms Will be Measured by the Patient Health Questionnaire-2 (PHQ-2).
Description: Participants' risk of depression will be measured by the Patient Health Questionnaire-2 (PHQ-2). This is a 2 item scale (with a 4 level Likert scale ranging from "Not at all" to "Nearly everyday") and the score ranges from 0-6, with a higher score indicating higher risk of depression.
Time Frame: 8 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention - Dating Application Topic | Control - Health and Exercise Topic
Number analyzed (Participants) | 290 | 288
Score on a scale | 4.21 (1.46) | 4.05 (1.33)
Statistical Analysis 1: Comparison: Intervention - Dating Application Topic vs Control - Health and Exercise Topic; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: None applicable
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03685643/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03685643/SAP_001.pdf